CLINICAL TRIAL: NCT00601523
Title: Long-term Safety Study of Open-label Pramipexole Extended Release (ER) in Patients With Early Parkinson´s Disease (PD).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 248.633; 2007-004234-16 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Results first posted 2011-08-25 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

ARMS (2):
- Pramipexole (Active Comparator): Patient to receive Pramipexole ER 0.375-4.5 mg tabl form daily
  Interventions: Drug: Pramipexole
- Placebo (Placebo Comparator): Patient to receive placebo tablets identical to Pramipexole ER tablets. Only during transfer phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Patient to receive placebo tablets identical to Pramipexole ER tablets. Only during transfer phase.
  Arms: Placebo
Drug: Pramipexole — ER 0.375-4,5 mg
  Arms: Pramipexole

SUMMARY:
The general aim of this study is to obtain long-term safety and tolerability data on pramipexole ER, in daily doses from 0.375mg to 4.5mg once daily (q.d), in patients who have previously completed a pramipexole double-blind study in early PD (248.524(NCT00479401) or 248.636(NCT00558025) trial).

ELIGIBILITY:
Inclusion criteria:

1. Completion of the double-blind trial 248.524 or 248.636
2. Male or female patient with early idiopathic Parkinson´s disease (PD), and with a Modified Hoehn and Yahr stage of I to III.
3. Patient willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
4. Signed informed consent obtained before any study procedures are carried out (in accordance with International Conference on Harmonisation (ICH) - Good Clinical Practice (GCP) guidelines and local legislation).

Exclusion criteria:

1. Patients prematurely withdrawn from the double-blind trials 248.524 or 248.636.
2. Atypical parkinsonian syndromes due to drugs,metabolic disorders, encephalitis or degenerative diseases.
3. Any psychiatric disorder according to Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV) criteria that could prevent compliance or completion of the study and/or put the patient at risk if he/she takes part in the study.4.History of psychosis, except history of drug induced hallucinations.

5. Clinically significant electrocardiogram (ECG) abnormalities at baseline. 6.Clinically significant hypotension 7.Malignant melanoma or history of previously treated malignant melanoma. 8.Any other clinically significant disease, that could put the patient at risk or could prevent compliance or completion of the study. 9. Pregnancy or breast-feeding.

10. Sexually active female of childbearing potential not using a medically approved method of birth control for at least one month prior to the baseline and throughout the study.11 Serum levels of aspartate aminotransferase (AST) (SGOT), alanine aminotransferase (ALT) (SGPT), alkaline phosphatase or bilirubin > 2 upper limit of normal (ULN) at baseline 12. Patients with a creatinine clearance < 50 mL/min (estimated by the Cockcroft and Gault formula). 13. Motor complications under levodopa therapy (e.g. on-off phenomena, dyskinesia) at baseline.

14. Any medication (including intra-muscular formulations) with central dopaminergic antagonist activity within 4 weeks prior to the baseline visit. 15.Any of the following drugs within 4 weeks prior to baseline: methylphenidate, cinnarizine, amphetamines. 16. Flunarizine within 3 months prior to baseline.

17. Known hypersensitivity to pramipexole or its excipients. 18. Drug abuse (including alcohol), according to investigator´s judgement, within 2 years prior to baseline.

19. Participation in investigational drug studies other than trials 248.524 and 248.636 or use of other investigational drug within one month or five times the half-life of the investigational drug prior to baseline.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (119):
- United States (10):
  - 248.633.01004 Boehringer Ingelheim Investigational Site, Sun City, Arizona
  - 248.633.01018 Boehringer Ingelheim Investigational Site, Tempe, Arizona
  - 248.633.01016 Boehringer Ingelheim Investigational Site, La Jolla, California
  - 248.633.01013 Boehringer Ingelheim Investigational Site, Oxnard, California
  - 248.633.01008 Boehringer Ingelheim Investigational Site, Danbury, Connecticut
  - 248.633.01010 Boehringer Ingelheim Investigational Site, Boca Raton, Florida
  - 248.633.01012 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 248.633.01001 Boehringer Ingelheim Investigational Site, Kansas City, Kansas
  - 248.633.01005 Boehringer Ingelheim Investigational Site, Commack, New York
  - 248.633.01009 Boehringer Ingelheim Investigational Site, Burlington, Vermont
- Austria (2):
  - 248.633.43001 Boehringer Ingelheim Investigational Site, Innsbruck
  - 248.633.43004 Boehringer Ingelheim Investigational Site, Vienna
- Czechia (4):
  - 248.633.42004 Boehringer Ingelheim Investigational Site, Olomouc
  - 248.633.42003 Boehringer Ingelheim Investigational Site, Pardubice
  - 248.633.42001 Boehringer Ingelheim Investigational Site, Prague
  - 248.633.42002 Boehringer Ingelheim Investigational Site, Rychnov nad Kněžnou
- Finland (3):
  - 248.633.35803 Boehringer Ingelheim Investigational Site, Hyvinkää
  - 248.633.35801 Boehringer Ingelheim Investigational Site, Oulu
  - 248.633.35802 Boehringer Ingelheim Investigational Site, Tampere
- France (32):
  - 248.633.3303A Boehringer Ingelheim Investigational Site, Aix-en-Provence
  - 248.633.3303B Boehringer Ingelheim Investigational Site, Aix-en-Provence
  - 248.633.3303C Boehringer Ingelheim Investigational Site, Aix-en-Provence
  - 248.633.3309A Boehringer Ingelheim Investigational Site, Clermont-Ferrand
  - 248.633.3309B Boehringer Ingelheim Investigational Site, Clermont-Ferrand
  - 248.633.3305A Boehringer Ingelheim Investigational Site, Créteil
  - 248.633.3305B Boehringer Ingelheim Investigational Site, Créteil
  - 248.633.3313A Boehringer Ingelheim Investigational Site, Dijon
  - 248.633.3304A Boehringer Ingelheim Investigational Site, Évreux
  - 248.633.3308A Boehringer Ingelheim Investigational Site, Lille
  - 248.633.3308B Boehringer Ingelheim Investigational Site, Lille
  - 248.633.3308C Boehringer Ingelheim Investigational Site, Lille
  - 248.633.3308D Boehringer Ingelheim Investigational Site, Lille
  - 248.633.3308E Boehringer Ingelheim Investigational Site, Lille
  - 248.633.3302A Boehringer Ingelheim Investigational Site, Marseille
  - 248.633.3302B Boehringer Ingelheim Investigational Site, Marseille
  - 248.633.3302C Boehringer Ingelheim Investigational Site, Marseille
  - 248.633.3306B Boehringer Ingelheim Investigational Site, Montpellier
  - 248.633.3306C Boehringer Ingelheim Investigational Site, Montpellier
  - 248.633.3306D Boehringer Ingelheim Investigational Site, Montpellier
  - 248.633.3306F Boehringer Ingelheim Investigational Site, Montpellier
  - 248.633.3306A Boehringer Ingelheim Investigational Site, Montpellier Cédex 5
  - 248.633.3312A Boehringer Ingelheim Investigational Site, Rouen
  - 248.633.3312B Boehringer Ingelheim Investigational Site, Rouen
  - 248.633.3311A Boehringer Ingelheim Investigational Site, Strasbourg
  - 248.633.3311B Boehringer Ingelheim Investigational Site, Strasbourg
  - 248.633.3301A Boehringer Ingelheim Investigational Site, Toulouse
  - 248.633.3301B Boehringer Ingelheim Investigational Site, Toulouse
  - 248.633.3301C Boehringer Ingelheim Investigational Site, Toulouse
  - 248.633.3301D Boehringer Ingelheim Investigational Site, Toulouse
  - 248.633.3301F Boehringer Ingelheim Investigational Site, Toulouse
  - 248.633.3301G Boehringer Ingelheim Investigational Site, Toulouse
- Germany (15):
  - 248.633.49009 Boehringer Ingelheim Investigational Site, Achim Bei Bremen
  - 248.633.49002 Boehringer Ingelheim Investigational Site, Berlin
  - 248.633.49004 Boehringer Ingelheim Investigational Site, Berlin
  - 248.633.49018 Boehringer Ingelheim Investigational Site, Berlin
  - 248.633.49019 Boehringer Ingelheim Investigational Site, Berlin
  - 248.633.49005 Boehringer Ingelheim Investigational Site, Bochum
  - 248.633.49016 Boehringer Ingelheim Investigational Site, Bochum
  - 248.633.49007 Boehringer Ingelheim Investigational Site, Dresden
  - 248.633.49011 Boehringer Ingelheim Investigational Site, Gera
  - 248.633.49017 Boehringer Ingelheim Investigational Site, Karlsruhe
  - 248.633.49001 Boehringer Ingelheim Investigational Site, Kassel
  - 248.633.49012 Boehringer Ingelheim Investigational Site, Leipzig
  - 248.633.49013 Boehringer Ingelheim Investigational Site, Marburg
  - 248.633.49003 Boehringer Ingelheim Investigational Site, Steglitz
  - 248.633.49015 Boehringer Ingelheim Investigational Site, Unterhaching
- Hungary (8):
  - 248.633.36007 Boehringer Ingelheim Investigational Site, Eger
  - 248.633.36005 Boehringer Ingelheim Investigational Site, Győr
  - 248.633.36008 Boehringer Ingelheim Investigational Site, Miskolc
  - 248.633.36004 Boehringer Ingelheim Investigational Site, Sopron
  - 248.633.36001 Boehringer Ingelheim Investigational Site, Szeged
  - 248.633.36006 Boehringer Ingelheim Investigational Site, Szeged
  - 248.633.36003 Boehringer Ingelheim Investigational Site, Szombathely
  - 248.633.36002 Boehringer Ingelheim Investigational Site, Zalaegerszeg
- India (7):
  - 248.633.91002 Boehringer Ingelheim Investigational Site, Chennai
  - 248.633.91009 Boehringer Ingelheim Investigational Site, Hyderabad
  - 248.633.91001 Boehringer Ingelheim Investigational Site, Karnataka
  - 248.633.91005 Boehringer Ingelheim Investigational Site, Maharashtra
  - 248.633.91007 Boehringer Ingelheim Investigational Site, Maharashtra
  - 248.633.91004 Boehringer Ingelheim Investigational Site, New Delhi
  - 248.633.91011 Boehringer Ingelheim Investigational Site, Pune
- Japan (15):
  - 248.633.81010 Boehringer Ingelheim Investigational Site, Aomori, Aomori
  - 248.633.81001 Boehringer Ingelheim Investigational Site, Bunkyo-ku, Tokyo
  - 248.633.81005 Boehringer Ingelheim Investigational Site, Fuchu, Tokyo
  - 248.633.81011 Boehringer Ingelheim Investigational Site, Fujisawa, Kanagawa
  - 248.633.81013 Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - 248.633.81015 Boehringer Ingelheim Investigational Site, Iwamizawa,Hokkaido
  - 248.633.81003 Boehringer Ingelheim Investigational Site, Kodaira, Tokyo
  - 248.633.81014 Boehringer Ingelheim Investigational Site, Kyoto, Kyoto
  - 248.633.81009 Boehringer Ingelheim Investigational Site, Morioka, Iwate
  - 248.633.81008 Boehringer Ingelheim Investigational Site, Okayama, Okayama
  - 248.633.81006 Boehringer Ingelheim Investigational Site, Ota-ku, Tokyo
  - 248.633.81004 Boehringer Ingelheim Investigational Site, Sagamihara, Kanagawa
  - 248.633.81007 Boehringer Ingelheim Investigational Site, Shimogyo-ku, Kyoto, Kyoto
  - 248.633.81012 Boehringer Ingelheim Investigational Site, Shiroishi, Miyagi
  - 248.633.81002 Boehringer Ingelheim Investigational Site, Takamatsu, Kagawa
- 248.633.60004 Boehringer Ingelheim Investigational Site, Kuala Terengganu, Malaysia
- Netherlands (5):
  - 248.633.31002 Boehringer Ingelheim Investigational Site, Geldrop
  - 248.633.31003 Boehringer Ingelheim Investigational Site, Helmond
  - 248.633.31006 Boehringer Ingelheim Investigational Site, Maastricht
  - 248.633.31004 Boehringer Ingelheim Investigational Site, Nijmegen
  - 248.633.31001 Boehringer Ingelheim Investigational Site, Sittard-geleen
- Russia (5):
  - 248.633.07001 Boehringer Ingelheim Investigational Site, Moscow
  - 248.633.07002 Boehringer Ingelheim Investigational Site, Moscow
  - 248.633.07003 Boehringer Ingelheim Investigational Site, Moscow
  - 248.633.07004 Boehringer Ingelheim Investigational Site, Moscow
  - 248.633.07006 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Slovakia (2):
  - 248.633.42103 Boehringer Ingelheim Investigational Site, Dubnica nad Váhom
  - 248.633.42101 Boehringer Ingelheim Investigational Site, Trnava
- Taiwan (4):
  - 248.633.88603 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 248.633.88605 Boehringer Ingelheim Investigational Site, Taichung
  - 248.633.88601 Boehringer Ingelheim Investigational Site, Taipei
  - 248.633.88602 Boehringer Ingelheim Investigational Site, Taoyuan District
- Ukraine (6):
  - 248.633.38005 Boehringer Ingelheim Investigational Site, Kiev
  - 248.633.38001 Boehringer Ingelheim Investigational Site, Lviv
  - 248.633.38002 Boehringer Ingelheim Investigational Site, Uzhhorod
  - 248.633.38003 Boehringer Ingelheim Investigational Site, Vinnytzya
  - 248.633.38004 Boehringer Ingelheim Investigational Site, Zaporizhzhya
  - 248.633.38006 Boehringer Ingelheim Investigational Site, Zaporizhzhya

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients From 248.524: Pramipexole ER 0.375-4.5 mg. Stratified cohort of patients who had previously completed 248.524 (NCT00479401) and previously received Pramipexole Extended Release (PPX ER), Pramipexole Immediate Release (PPX IR), or Placebo.
- Patients From 248.636: Pramipexole ER 0.375-4.5 mg. Stratified cohort of patients who had previously completed 248.636 (NCT00558025) and previously received Pramipexole Extended Release (PPX ER), Pramipexole Immediate Release (PPX IR), or Placebo.
Period: Overall Study
Arm/Group | Patients From 248.524 | Patients From 248.636
Started | 368 | 143
Completed | 291 | 117
Not Completed | 77 | 26
Not completed — Adverse Event | 42 | 14
Not completed — Lack of Efficacy | 3 | 0
Not completed — Protocol Violation | 5 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 18 | 9
Not completed — Other | 9 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set, all patients randomized and received treatment
Groups:
- Patients From 248.524: Patients who had previously completed 248.524 (NCT00479401)
- Patients From 248.636: Patients who had previously completed 248.636 (NCT00558025)
- Total: Total of all reporting groups
Arm/Group | Patients From 248.524 | Patients From 248.636 | Total
Number analyzed (Participants) | 368 | 143 | 511
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.2 (9.2) | 64.0 (9.0) | 62.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164 | 62 | 226
  Male | 204 | 81 | 285

OUTCOME MEASURES:

1. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) II+III Total Score: Change From Baseline
Description: UPDRS II+III ranging from 0 (normal) to 160 (severe). UPDRS part II measures activities of daily living, part III measures motor symptoms
Time Frame: Open Label (OL) baseline and week 80 (patients from 248.524) or week 72 (patients from 248.636)
Population: Patients from Full Analysis Set (FAS included all patients who received at least one dose of study medication and had at least one post-baseline efficacy assessment) and who had values for UPDRS II+III at week 80 (patients from 248.524) or at week 72 (patients from 248.636)
Measure: Mean (Standard Deviation); unit: Units of scale
Arm/Group | Patients From 248.524 | Patients From 248.636
Number analyzed (Participants) | 290 | 113
Units of scale | 2.2 (9.5) | 1.5 (7.7)

2. Secondary Outcome: Number of Patients With UPDRS II+III Response From OL Baseline at Week 80 (Patients From 248.524) or Week 72 (Patients From 248.636)
Description: A response means an improvement of >=20% from OL baseline. UPDRS II+III ranging from 0 (normal) to 160 (severe). UPDRS part II measures activities of daily living, part III measures motor symptoms
Time Frame: OL Baseline and week 80 (patients from 248.524) or week 72 (patients from 248.636)
Population: as for outcome 1
Measure: Number; unit: Patients
Arm/Group | Patients From 248.524 | Patients From 248.636
Number analyzed (Participants) | 289 | 113
Patients | 73 | 27

3. Secondary Outcome: UPDRS I Total Score: Change From OL Baseline
Description: UPDRS I ranging from 0 (normal) to 16 (severe), measures Mentation, Behavior and Mood
Time Frame: OL baseline and week 80 (patients from 248.524) or week 72 (patients from 248.636)
Population: Patients from FAS and who had values for UPDRS I at week 80 (patients from 248.524) or at week 72 (patients from 248.636)
Measure: Mean (Standard Deviation); unit: Units of scale
Arm/Group | Patients From 248.524 | Patients From 248.636
Number analyzed (Participants) | 287 | 111
Units of scale | 0.3 (1.0) | 0.1 (1.3)

4. Secondary Outcome: UPDRS II Total Score: Change From OL Baseline
Description: UPDRS II ranging from 0 (normal) to 52 (severe), measures activity of daily living.
Time Frame: OL baseline and week 80 (patients from 248.524) or week 72 (patients from 248.636)
Population: Patients from FAS and who had values for UPDRS II at week 80 (patients from 248.524) or at week 72 (patients from 248.636)
Measure: Mean (Standard Deviation); unit: Units of scale
Arm/Group | Patients From 248.524 | Patients From 248.636
Number analyzed (Participants) | 290 | 113
Units of scale | 1.0 (3.2) | 0.6 (3.5)

5. Secondary Outcome: UPDRS III Total Score: Change From OL Baseline
Description: UPDRS III ranging from 0 (normal) to 108 (severe) measures motor symptoms
Time Frame: OL baseline and week 80 (patients from 248.524) or week 72 (patients from 248.636)
Population: Patients from FAS and who had values for UPDRS III at week 80 (patients from 248.524) or at week 72 (patients from 248.636)
Measure: Mean (Standard Deviation); unit: Units of scale
Arm/Group | Patients From 248.524 | Patients From 248.636
Number analyzed (Participants) | 290 | 113
Units of scale | 1.1 (7.2) | 0.9 (5.6)

6. Secondary Outcome: Response in Clinical Global Impression of Improvement (CGI-I)
Description: Clinicians evaluation in a rating scale of 7 steps, 1 meaning very much improved to 7 meaning very much worse. For patients previously treated with Placebo, all patients with at least "much improved" were considered as responders. For patients previously treated with Pramipexole ER or Immediate Release (IR), all patients with no change to very much improved were considered as responders
Time Frame: OL Baseline and week 32 (patients from 248.524) or week 24 (patients from 248.636)
Population: Patients from FAS and who had values for for CGI-I at week 32 (patients from 248.524) or at week 24 (patients from 248.636)
Measure: Number; unit: Patients
Arm/Group | Patients From 248.524 | Patients From 248.636
Number analyzed (Participants) | 336 | 133
Patients | 284 | 108

7. Secondary Outcome: Response in Patient Global Impression of Improvement (PGI-I)
Description: Patient rated evaluation of the PD symptoms on a rating scale of 7 steps, 1 meaning very much better to 7 meaning very much worse. For patients previously treated with Placebo, all patients with at least "much better" were considered as responders. For patients previously treated with pramipexole (PPX) ER or IR, all patients with no change to very much better were considered as responders
Time Frame: OL Baseline and week 32 (patients from 248.524) or week 24 (patients from 248.636)
Population: Patients from FAS and who had values for for PGI-I at week 32 (patients from 248.524) or at week 24 (patients from 248.636)
Measure: Number; unit: Patients
Arm/Group | Patients From 248.524 | Patients From 248.636
Number analyzed (Participants) | 336 | 133
Patients | 265 | 111

8. Secondary Outcome: Parkinson Fatigue Scale (PFS-16) : Change From OL Baseline
Description: PFS-16 ranging from 16 (better perceived health status) to 80 (severe symptoms of the disease) measuring aspects of fatigue that are relevant to patients with PD.
Time Frame: OL baseline and week 80 (patients from 248.524) or week 72 (patients from 248.636)
Population: Patients from FAS and who had values for PFS-16 at week 80 (patients from 248.524) or at week 72 (patients from 248.636)
Measure: Mean (Standard Deviation); unit: Units of scale
Arm/Group | Patients From 248.524 | Patients From 248.636
Number analyzed (Participants) | 303 | 110
Units of scale | 2.0 (12.5) | 2.2 (9.8)

9. Secondary Outcome: Number of Patients Introducing L-Dopa Medication in OL Trial
Description: Number of patients requiring Levodopa supplementation during the study
Time Frame: 80 weeks (patients from 248.524) or 72 weeks (patients from 248.636)
Population: Patients from FAS
Measure: Number; unit: Patients
Arm/Group | Patients From 248.524 | Patients From 248.636
Number analyzed (Participants) | 367 | 138
Patients
  No | 320 | 117
  Yes | 47 | 21

10. Secondary Outcome: L-Dopa Dose: Change From OL Baseline
Description: Change from open-label baseline in Levodopa dose
Time Frame: OL baseline and week 80 (patients from 248.524) or week 72 (patients from 248.636)
Population: Patients from FAS and with L-Dopa at OL baseline and at week 80 (patients from 248.524) or week 72 (patients from 248.636)
Measure: Number; unit: Patients
Arm/Group | Patients From 248.524 | Patients From 248.636
Number analyzed (Participants) | 32 | 64
Patients
  Decrease | 4 | 0
  Increase | 9 | 23
  No change | 19 | 41

11. Secondary Outcome: Pramipexole Doses Respectively After 80 Weeks Compared to Pramipexole Doses at Week 8 for Previously 248.524 Patients and After 72 Weeks Compared to Pramipexole Doses at Week 0 for Previously 248.636 Patients
Description: Change from open-label baseline in Levodopa dose over the final 72 weeks of open-label assessment
Time Frame: Week 8 and week 80 (patients from 248.524) or week 0 and week 72 (patients from 248.636)
Population: Patients from Treated Set (defined as all patients who were dispensed study drug and were documented to have at least one dose of investigational treatment) and treated until week 80 (patients from 248.524) or week 72 (patients from 248.636)
Measure: Number; unit: Patients
Arm/Group | Patients From 248.524 | Patients From 248.636
Number analyzed (Participants) | 339 | 126
Patients
  Decrease | 101 | 9
  Increase | 82 | 44
  No change | 156 | 73

12. Primary Outcome: Percentage of Patients With Adverse Events, Adverse Drug Reactions, Serious Adverse Events
Description: The aim of this study was to obtain long-term safety and tolerability data on pramipexole ER, in patients who have previously completed a pramipexole double blind study in early PD (248.524 (NCT00479401) or 248.636 (NCT00558025)). Therefore these items were considered as a safety evaluation
Time Frame: 80 weeks (patients from 248.524) or 72 weeks (patients from 248.636)
Population: Patients from Treated Set (defined as all patients who were dispensed study drug and were documented to have at least one dose of investigational treatment)
Measure: Number; unit: Percentage of participants
Arm/Group | Patients From 248.524 | Patients From 248.636
Number analyzed (Participants) | 368 | 143
Percentage of participants
  Percentage of Patients with Adverse Events | 84.5 | 76.2
  Percentage of Patients with Adverse Drug Reactions | 45.7 | 23.1
  Percentage of Patients with Serious Adverse Events | 14.4 | 14.7

13. Secondary Outcome: Patient Preference Regarding Treatment Dosing
Description: Patients were surveyed on their preference for Once Daily dosing versus Three Times Daily dosing
Time Frame: 80 weeks (patients from 248.524) or 72 weeks (patients from 248.636)
Population: Patients from Full Analysis Set (FAS included all patients who received at least one dose of study medication and had at least one post-baseline efficacy assessment)
Measure: Number; unit: participants
Arm/Group | Patients From 248.524 | Patients From 248.636
Number analyzed (Participants) | 367 | 138
participants
  Prefer Once Daily dosing | 275 | 78
  Prefer 3 Times Daily dosing | 9 | 1
  No Preference | 7 | 4
  Missing | 76 | 55

14. Secondary Outcome: Patient Rating of Convenience of Treatment Dosing
Description: Patients were surveyed on the convenience of Once Daily dosing versus Three Times Daily dosing
Time Frame: 80 weeks (patients from 248.524) or 72 weeks (patients from 248.636)
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Patients From 248.524 | Patients From 248.636
Number analyzed (Participants) | 367 | 138
participants
  Once Daily much more convenient | 196 | 59
  Once Daily more convenient | 79 | 19
  3 Times Daily much more convenient | 2 | 0
  3 Times Daily more convenient | 6 | 1
  No difference in preference | 7 | 4
  Missing | 77 | 55

ADVERSE EVENTS:
Time Frame: Up to 80 weeks for patients from 248.524, Up to 72 weeks for patients from 248.636
Arm/Group | Patients From 248.524 | Patients From 248.636
Serious Adverse Events (participants affected / at risk) | 53/368 | 21/143
Other Adverse Events (participants affected / at risk) | 214/368 | 62/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients From 248.524 (N=368) | Patients From 248.636 (N=143)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 4 | 1
Myocardial rupture (Cardiac disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Drowning (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Borrelia infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Prostatic abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 3
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Arthroscopy (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cervical root pain (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
On and off phenomenon (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 2 | 2
Sciatica (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 2 | 1
Psychotic disorder (Psychiatric disorders) | 2 | 0
Sleep attacks (Psychiatric disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Hydroureter (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1
Cystocele (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Varicose vein (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients From 248.524 (N=368) | Patients From 248.636 (N=143)
Cataract (Eye disorders) | 25 | 7
Constipation (Gastrointestinal disorders) | 15 | 9
Nausea (Gastrointestinal disorders) | 37 | 10
Oedema peripheral (General disorders) | 45 | 15
Nasopharyngitis (Infections and infestations) | 29 | 8
Fall (Injury, poisoning and procedural complications) | 20 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 40 | 13
Dizziness (Nervous system disorders) | 32 | 3
Parkinson's disease (Nervous system disorders) | 7 | 10
Somnolence (Nervous system disorders) | 67 | 10
Hallucination (Psychiatric disorders) | 8 | 8
Insomnia (Psychiatric disorders) | 19 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.